CLINICAL TRIAL: NCT01538537
Title: Phase I Dose Escalation Study of ON 01910.Na by 3-day Continuous Infusion in Patients With Advanced Cancer
Brief Title: Safety of ON 01910.Na as a 3-day Infusion in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-02
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Advanced Cancer; Solid Tumors; Cancer; Neoplasms
Keywords: ON 01910.Na; rigosertib Sodium; rigosertib
MeSH Terms: conditions — Neoplasms | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rigosertib sodium — ON 01910.Na will be supplied as a sterile, concentrated solution (75 mg/ml) in labeled, sealed glass vials. ON 01910.Na concentrated solution (75 mg/ml) must be diluted before intravenous administration. The starting dose will be 50 mg/m2 over 24 hour infusion daily for 3 days. A fresh infusion must be prepared for each day of the 3-day continuous infusion. This 3-day continuous treatment followed by 11 days without administration of study drug will constitute 1 Cycle. Cycles can be repeated every 2 weeks. The dosing of ON 01910.Na will be based on body surface area (BSA). In the absence of toxicity that would cause accelerated dose escalation to cease, drug doses are planned to escalate every 3 weeks.
  Other Names: ON 01910.Na Concentrate; ON 01910.Na; rigosertib

SUMMARY:
The primary objective of this study is to determine the largest dose of ON 01910.Na (rigosertib sodium) that can be given safely as a 3-day continuous infusion once every 2 weeks (2-week cycle) in patients with advanced cancer.

DETAILED DESCRIPTION:
This was an open-label, single-center, dose-escalating Phase I study to determine the Dose-Limiting Toxicities (DLTs) and Recommended Phase 2 Dose (RPTD) of ON 01910.Na (rigosertib sodium) administered as a 3 day continuous intravenous (CIV) infusion every 2 weeks (2-week cycles) to up to 28 patients with advanced cancer (12 to 16 in the dose escalation phase and up to 12 additional patients in the dose confirmation phase). The dosing of rigosertib was based on body surface area (BSA), with a starting dose of 50 mg/m2/24 hour for 3 consecutive days.

In the absence of toxicity after at least a 3-week observation period, rigosertib doses were escalated following a Fibonacci scheme with an initial accelerated dose-escalation phase in which 1-patient cohorts received rigosertib for 3 weeks until drug-related Grade 2 toxicity (according to Common Toxicity Criteria for Adverse Events [CTCAE] v.3), excluding alopecia, occurred, at which time 2 additional patients were added to subsequent cohorts. If none of the 3 patients in the cohort experienced DLTs, the dose was escalated by a half-Fibonacci step. If a DLT was seen in the first patient of a cohort, dosing went back a half-step. The next dose level occurred if no DLT was reported in the 3 patients or if no more than 1 DLT occurred in an expanded cohort of 6 patients. If a DLT was seen in 1 of the 3 patients, 3 additional patients were enrolled in the cohort. If DLTs were seen in 2 of 6 patients in a cohort, dose escalation was stopped.

Once the maximum administered dose (MAD) was attained and the RPTD was determined, the dose escalation phase was considered complete. Up to 12 additional patients with histologically confirmed malignant tumors were tested at the RPTD dose to confirm its appropriateness.

Secondary objectives were to determine the qualitative and quantitative toxicity and reversibility of toxicity of rigosertib administered in this fashion; to investigate the clinical pharmacology of rigosertib when administered in this fashion, including plasma pharmacokinetics at each dose level; to confirm the appropriateness of the RPTD; to document any observed antitumor activity of rigosertib; and, to evaluate the biological effect of rigosertib in biomarkers in serum and/or peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* At least 4 weeks since the last dose of other potentially myelosuppressive treatment (at least 6 weeks since last dose of nitrosoureas or mitomycin C) and recovery from manifestations of reversible drug toxicity (except alopecia, stable residual neuropathy, and residual hand and foot syndrome). Among patients with prior doxorubicin chemotherapy, only those with no more than 450 mg/m2 of the drug will be entered. It must be at least 4 weeks since prior chemotherapy or radiation therapy, 6 weeks if the last regimen included nitrosoureas or mitomycin C.
* Patients with prior radiotherapy are eligible provided that a minimum of 4 weeks have passed and that the maximal area of hematopoietic active bone marrow treated was less than 25%.
* ECOG performance status < 2.
* Hgb > 10 gm/dl
* WBC > 4,000 per microliter
* Absolute neutrophil count > 1,500 per microliter
* Platelets >100,000 per microliter
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) values within limits defined by Protocol
* Creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Women of child-bearing potential and men must agree to use adequate contraception.
* Ability to understand and the willingness to sign a written informed consent document.

Inclusion Criteria - Dose Confirmation Phase Same inclusion criteria as in the Dose Escalation phase described above, except Patients must have an ECOG performance of 0 or 1.

Exclusion Criteria:

* Patients who have had recent major surgery (within the past 14 days), chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (except alopecia, stable residual neuropathy, and residual hand and foot syndrome) due to previously administered agents.
* Patients may not be receiving any other investigational agents or concurrent chemotherapy, radiotherapy, hormonal treatments, or immunotherapy while on study.
* Patients with known or clinical evidence of central nervous system metastasis, except brain metastases that have been previously removed or irradiated and currently have no clinical impact.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ON 01910.Na.
* The patient should have no major 3rd space fluid, ascites requiring active medical management including paracentesis, peripheral bilateral edema, or hyponatremia (serum sodium value less than 134 Meq/L).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, bleeding, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women are excluded from this study.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-08; Primary Completion 2010-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of dose limiting toxicities (DLTs) | 28 days after start of first administration of ON 01910.Na
  DLTs are defined as:
  * Grade 3 non-hematological toxicity other than nausea, vomiting, diarrhea, fever, stomatitis, esophagitis/dysphagia.
  * Grade 3 nausea and vomiting uncontrolled by antiemetics; Grade 3 diarrhea uncontrolled by antidiarrheal agents; Grade 3 drug-induced fever uncontrolled by antipyretics.
  * Grade 3 stomatitis and/or esophagitis/dysphagia lasting >3 days.
  * Grade 4 neutropenia or thrombocytopenia lasting >5 days.
  * Episode of neutropenic fever, as defined in Protocol.
  * Failure to recover neutrophils (>1,500 per microliter) or platelets (>75,000 per microliter) by day 28.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | 30 days after last infusion of study drug
  All adverse events (except grade 1 and 2 laboratory abnormalities that do not require an intervention), regardless of causal relationship, are recorded in the case report form and source documentation.
Severity of Adverse Events | 30 days after last infusion of study drug
  Severity of AEs are determined according to the NCI Common Terminology Criteria for Adverse Events, Version 3.0.
Relationship of Adverse Events (AEs) to Study Treatment | 30 days after last infusion of study drug
  Relationship assessed as Not related, Unlikely, Possibly, Probably, or, Definitely according to Guidance in Appendix II of Protocol.
Concentration of ON 01910.Na in plasma versus time | Up to 72 hours after end of infusion of study drug in Cycles 1 and 4
  Blood samples for subsequent preparation of plasma and determination of concentration of ON 01910.Na will be collected at pre-dose at 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 72 hr (10 min, prior to completion of infusion). After the completion of the infusion, samples will be collected at 10 min, 20 min, 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 24 hr, 48 hr, and 72 hr.
Change in size of target lesions recorded at baseline | 30 days after last infusion of study drug
  The same method of assessment for each identified and recorded lesion will be used at baseline and each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Takao Ohnuma, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Ohnuma T, Lehrer D, Ren C, Cho SY, Maniar M, Silverman L, Sung M, Gretz HF 3rd, Benisovich V, Navada S, Akahoho E, Wilck E, Taft DR, Roboz J, Wilhelm F, Holland JF. Phase 1 study of intravenous rigosertib (ON 01910.Na), a novel benzyl styryl sulfone structure producing G2/M arrest and apoptosis, in adult patients with advanced cancer. Am J Cancer Res. 2013 Jun 20;3(3):323-38. Print 2013. PMID 23841031
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.